CLINICAL TRIAL: NCT05773456
Title: Iodine Status at Several Time Points During 48 Hours After Intake of Sushi and Seaweed Salad- a Randomized Crossover Trial
Brief Title: Iodine Status After Intake of Sushi and Seaweed Salad
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bergen (Other)
Collaborators: Institute of Marine Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 232247
Record Dates: First submitted 2023-03-06; First posted 2023-03-17 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-01

CONDITIONS: Iodine Deficiency
Keywords: seaweed; bioavailability; iodine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sushi and wakame salad (Experimental): 231 microgram of iodine per serving
  Interventions: Other: Sushi and wakame salad
- Potassium iodide supplement (Active Comparator): 225 microgram of iodine per tablet
  Interventions: Other: Sushi and wakame salad

INTERVENTIONS:
Other: Sushi and wakame salad — One serving of mixed sushi and wakame salad

SUMMARY:
Seaweed is becoming increasingly popular in the Western part of the world, especially sushi wrapped in nori and seaweed salad, also called wakame. There are limited data on the iodine content of different seaweed products in the Norwegian Food composition table. Furthermore, there is limited available research regarding in vivo bioavailability of iodine from seaweeds. The objective of this study is to assess whether iodine from a sushi meal (with nori, Porphyra spp), and a wakame salad (Undaria pinnatifida) has similar bioavailability as a potassium iodide reference supplement of similar iodine content.

ELIGIBILITY:
Inclusion Criteria:

* healthy women aged 18 to 40 years

Exclusion Criteria:

* pregnant or lactating
* known thyroid disease or thyroid autoimmunity,
* planning to conceive,
* known kidney problems or kidney disease.
* women with coeliac disease could not participate due to possible gluten exposure from the wakame salad

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2021-08-10 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
Urinary iodine concentration during 48 hours | 48 hours
  Urinary iodine concentration after ingestion of the intervention/supplement during 48 hours by fixed time-intervals
Bio-availability of iodine in the intervention/supplement | 48 hours
  Calculation of the bio-availability of iodine in the intervention/supplement

CONTACTS AND LOCATIONS:
Overall Officials: Inger Aakre, PhD, Principal Investigator — Institute of Marine Research
Locations (1):
- University of Bergen, Bergen, Norway

IPD SHARING:
Plan to Share IPD: No